CLINICAL TRIAL: NCT03277963
Title: Perception of Pain During Obstructive Sleep Apnea Syndrome in Obese Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CHU-348; 2008-A01045-50 (Other: 2008-A01045-50)
Record Dates: First submitted 2017-09-04; First posted 2017-09-11 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Obstructive Sleep Apnea Syndrome
Keywords: Obesity; Obstructive sleep apnea syndrome
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absence of sleep apnea syndrome (Active Comparator): Pain perception tests
  Interventions: Device: Pain perception tests (mechanical : VON FREY ELECTRONIQUE or electrical stimulus : PAIN MATCHER®)
- Presence of sleep apnea syndrome (Experimental): Pain perception tests and for severe sleep apnea syndrome, treatment by positive airway pressure (PPC) ventilation
  Interventions: Device: Pain perception tests (mechanical : VON FREY ELECTRONIQUE or electrical stimulus : PAIN MATCHER®)

INTERVENTIONS:
Device: Pain perception tests (mechanical : VON FREY ELECTRONIQUE or electrical stimulus : PAIN MATCHER®) — From a basal level causing no particular sensation, the mechanical or electrical stimulus is applied with a constant increasing rate of progression.

SUMMARY:
Obstructive sleep apnea syndrome (SAOS), very commonly associated with obesity, induces major disturbances in sleep architecture. The hypotheses in this work are twofold: on the one hand, the SAOS could generate pain perception disorders in a population already affected by the mechanical weight constraints, generating potentially painful complications, and on the other hand, the improvement of sleep provided by continuous positive airway pressure (PPC) ventilation could "normalize" the pain perception thresholds. It was shown an early rebound effect after treatment on increasing pain threshold in the healthy subject. We want to check it among obese patients with OSA in early and mid-term.

DETAILED DESCRIPTION:
In this controlled study, patients of both sexes over 18 years of age who are obese with a body mass index (BMI) of 30 will be included. They will benefit from a polygraphy to confirm or invalidate the presence of an obstructive sleep apnea syndrome (defined by an apnea-hypopnea index to 10). Patients will be tested for mechanical and electrical pain within one week of diagnosis. Among these patients, those with severe SAOS (IAH 30) warrant treatment with continuous positive airway pressure (usual procedure). They will be hospitalized for the implementation of this treatment (usual procedure) and subjected to mechanical and electrical pain tests on the second day after the treatment is put in place.

One month after the start of treatment, they will benefit from an ambulatory polygraph test (usual procedure) as well as mechanical and electrical pain tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age,
* male or female,
* obesity defined by a body mass index (BMI = weight in kg / height in m²) ≥ 30,
* free from acute or chronic painful pathology,
* free from any chronic analgesic treatment,
* free from any psychotropic treatment by benzodiazepine and / or tricyclic antidepressant,
* presence of obstructive sleep apnea syndrome (with apnea-hypopnea index (IAH) 10 per hour of sleep) among 60 patients,
* absence of obstructive sleep apnea syndrome (IAH <10 per hour of sleep) among 60 patients,
* person who signed the information and consent form,
* patients who have been screened for sleep apnea syndrome by Somnochek® negative (AHI <10 / h) in the last 6 months, provided that their weight is the same or lower at the time of inclusion,
* Somnochek® sleep apnea syndrome screening positive and severe for hospitalization (IAH> 30 / h) in the last 3 months, provided that their weight is the same or higher at the time of inclusion.

In addition, the 23 patients in the subgroup with severe OSA must meet the following criteria:

* presence of obstructive sleep apnea syndrome (with apnea-hypopnea index (IAH) 30 per hour of sleep) among 23 patients,
* acceptance of treatment with PCC,
* availability to come to the CHU for the control of pain threshold perception tests one month after the introduction of PPC treatment.

Exclusion Criteria:

* difficulties in understanding and speaking French,
* an alcohol abuse or dependence (DSM-IV),
* an abuse or dependence on illicit drugs (DSM-IV),
* an acute or chronic inflammatory pathology,
* a neuro-muscular pathology,
* clinical signs of right heart failure,
* an analgesic treatment,
* treatment with benzodiazepines and / or tricyclic antidepressants, a β-blocking treatment,
* Central sleep apnea,
* person who is absent from another study or who has received more than 4500 euros in the year following his participation in clinical studies,
* pregnant or nursing women,
* person under tutelage or deprived of his rights,
* refusal to sign the information and consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02-04 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
scales of pain | at day 1
  sensibility, detection, tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Magalie MIOLANNE-DEBOUIT, PH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France